CLINICAL TRIAL: NCT02116153
Title: Clinical Use of Mi-RNAs to Improve Specificity of High-sensitivity Troponin T in Symptomatic Patients Presenting to the ED
Brief Title: Mi-RNAs and Specificity of Hs-TnT in Symptomatic ED Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other)
Responsible Party: Principal Investigator, Professor Hugo Katus, Director, Department of Cardiology, University Hospital Heidelberg
Other Study IDs: UHHD-BM-003
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: Cardiac Troponin T; Micro-RNA; Sensitivity; Specificity
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Cardiomyopathy, Familial Restrictive, 3; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Biomarkers play a key role in the diagnostic workup of patients presenting to an emergency department (ED). European and American guidelines recommend cardiac Troponin (T or I) as the biomarker gold standard for the diagnosis of non-ST-elevation myocardial infarction (non-STEMI). Today, high-sensitivitiy assays are available and allow an early diagnosis of non-STEMI and the detection of troponin in individuals that would have been classified as unstable angina with former assays. As many patients are detected with elevated troponin values with the high sensitivity assays, specificity for non-STEMI has inevitably decreased. Micro-RNAs (mi-RNA) are new biomarkers with a wide spectrum of detectable conditions that allow specific identification of myocardial infarction. The aim of this study is to develop a biomarker protocol that combines the high sensitivity of cardiac Troponin T and the high specificity of mi-RNA profiles for early and safe identification of non-STEMI in ED patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency department ("chest pain unit"), Dept. of Cardiology, University Hospital Heidelberg
* Symptoms suggestive of ACS incl. chest pain, dyspnea, atypical pain
* Age >= 18 years
* Written informed consent

Exclusion Criteria:

* Mental disorders, dementia
* Pregnancy, breast feeding
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department with symptoms suggestive of acute coronary syndrome.
Sampling Method: Non-Probability Sample
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Death | 90 days

SECONDARY OUTCOMES:
Myocardial Infraction | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giannitsis, MD, Principal Investigator — University Hospital Heidelberg; Hugo A Katus, MD, Study Director — University Hospital Heidelberg

REFERENCES:
- [Derived] Biener M, Giannitsis E, Thum T, Bar C, Costa A, Andrzejewski T, Stoyanov KM, Vafaie M, Meder B, Katus HA, de Gonzalo-Calvo D, Mueller-Hennessen M. Diagnostic value of circulating microRNAs compared to high-sensitivity troponin T for the detection of non-ST-segment elevation myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2021 Aug 24;10(6):653-660. doi: 10.1093/ehjacc/zuaa034. PMID 33580779